CLINICAL TRIAL: NCT06290882
Title: Endoscopic Versus Robotic Myotomy for Treatment of Achalasia (ERMA Trial)
Brief Title: Endoscopic Versus Robotic Myotomy for Treatment of Achalasia
Acronym: ERMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Elisenda Garsot Savall, Head of Upper GI section, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERMA trial
Record Dates: First submitted 2024-01-25; First posted 2024-03-04 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Achalasia Cardia
Keywords: Achalasia; Robotic Heller Myotomy; Peroral Endoscopic Myotomy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Heller Myotomy. (Active Comparator): Patients with Achalasia, designated to receive a myotomy of the lower esophageal sphincter, who have been randomised into the Robotic Heller Myotomy group
  Interventions: Procedure: Robotic Heller Myotomy
- Peroral Endoscopic Myotomy. (Active Comparator): Patients with Achalasia, designated to receive a myotomy of the lower esophageal sphincter, who have been randomised into the Peroral Endoscopic Myotomy group
  Interventions: Procedure: Peroral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Robotic Heller Myotomy — Use five trocar technique with patient in the French position. Establish 12-15 mm Hg pneumoperitoneum. Divide phrenoesophageal ligament starting on the right and mobilize distal esophagus on the lateral and anterior side. Identify and spare anterior vagal nerve. Perform myotomy by dividing both muscle-layers extending at least 7 cm above gastroesophageal junction and 2 cm inferiorly over stomach. Measure myotomy length. Perform anterior fundoplication without mobilizeng fundus of the stomach by dividing short gastric vessels if not necessary. Suture fundus to both cut edges of myotomy, using non-resorbable material.
  Arms: Robotic Heller Myotomy.
Procedure: Peroral Endoscopic Myotomy — After lavage, measure gastro-esophageal junction (GEJ) in cm from mouth piece. Determine entry point 12-14cm above GEJ at the lesser curvature site, inject 10ml coloured saline, create entry point. Advance endoscope into the submucosa, dissect the submucosal tunnel up to 2-3cm into the cardia. Dissect the submucosa close to the muscularis and check endoluminally for the direction of the lesser curvature, sufficient extension onto the cardia and mucosal integrity. After tunnel completion flush with gentamycin and saline. Start myotomy from proximally to distally starting 4-5cm below the mucosal entry site; the inner circular muscle layer should be fully dissected especially at the cardia for good symptomatic results. It is vital that the mucosa of the tubular esophagus remains intact. Extend myotomy at least 2cm onto the cardia. After completion check for mucosal integrity and opening of the distal esophageal sphincter. Close the entry point with clips from distal to proximal.
  Arms: Peroral Endoscopic Myotomy.

SUMMARY:
Achalasia is a primary esophageal motor disorder of unknown etiology characterized by degeneration of the myenteric plexus, resulting in impaired relaxation of the esophagogastric junction (EGJ), along with loss of peristalsis in the esophageal body. The standard criteria for diagnosing achalasia is high-resolution esophageal manometry, which shows incomplete relaxation of the EGJ along with absence of esophageal body peristalsis. These anomalies usually cause dysphagia and regurgitation as the main symptoms of this pathology. Different treatment options have been described for this pathology, with pneumatic dilation (PD) and myotomy being considered first-line, whether surgical (laparoscopic Heller myotomy, LHM) or endoscopic (peroral endoscopic myotomy, POEM). The arrival of POEM as a less invasive alternative for the treatment of achalasia has revolutionized expectations to the point that it has become a routine procedure in many centers around the world. In recent years, a large amount of data examining the effectiveness of POEM have appeared, including several meta-analyses. The success rate of POEM in prospective cohorts has been greater than 90%. Two randomized studies have been published comparing POEM with LHM, providing a framework to evaluate the comparative efficacy and safety of these two interventions and to determine which should be first-line for the treatment of these patients. According to these data, it seems that the two procedures offer the same clinical results in the medium term. On the other hand, in recent years, there has been a growing expansion of the application of robot-assisted technology. Robotic Heller myotomy (RHM) has been proposed as an alternative minimally invasive approach to traditional laparoscopy with a lower complication rate. Based on the evidence, POEM and RHM could have comparable results in short term, but there is no clear certainty about the results in medium-long term. Likewise, there is a lack of studies that confirm postoperative reflux results in both procedures.

The purpose of the study is to evaluate the clinical and quality of life results of the RHM and compare them with the results of POEM in treatment of achalasia.

DETAILED DESCRIPTION:
Achalasia is a primary esophageal motor disorder of unknown etiology characterized by degeneration of the myenteric plexus, resulting in impaired relaxation of esophagogastric junction (EGJ), along with loss of peristalsis in the esophageal body. The standard criteria for diagnosing achalasia is high-resolution esophageal manometry, which shows incomplete relaxation of the EGJ along with absence of esophageal body peristalsis. These anomalies usually cause dysphagia and regurgitation as the main symptoms. Three subtypes of achalasia have been defined based on the findings of high-resolution manometry in the esophageal body: type I or classic achalasia with low intraesophageal pressure, type II with panesophageal pressurization, and type III with high-amplitude spastic contractions.

Different treatment options have been described for this pathology, with pneumatic dilation (PD) and myotomy being considered first-line, whether surgical (laparoscopic Heller myotomy, LHM) or endoscopic (peroral endoscopic myotomy, POEM). PD is the most frequently performed treatment worldwide with a reported long-term effectiveness between 50-93%, although it is generally a procedure that requires multiple sessions. On the other hand, LHM combined with an antireflux procedure is a treatment that, despite being more invasive, in most cases requires only one treatment session and offers success rates of 71% to 92%. POEM is a recently emerging procedure but with a success rate in prospective cohorts that sometimes exceeds 90%.

Multiple studies have shown that treatment outcomes depend on the subtype of achalasia. Based on available data, pneumatic dilation, laparoscopic Heller myotomy and POEM are believed to be effective for achalasia type I and II, while POEM has emerged as the preferred treatment for achalasia type III, which is believed to be related to the ability to perform a proximal extended myotomy. The arrival of POEM as a less invasive alternative for the treatment of achalasia has revolutionized expectations to the point that it has become a routine procedure in many centers around the world that use it for the treatment of any type of achalasia. In recent years, there is a large amount of data examining the effectiveness of POEM, including several meta-analyses. The success rate of POEM in prospective cohorts has been greater than 90% and has been maintained across all achalasia subtypes. Two randomized studies have been published comparing POEM with LHM, providing a framework to evaluate the comparative efficacy and safety of these two interventions and to determine which should be first-line for the treatment of these patients. With these data, it seems that the two procedures offer the same clinical results in the medium term.

However, the main issue that POEM faces is the presence of post-procedure reflux. The incidence of reflux disease seems to be significantly higher after POEM compared to LHM with fundoplication but the way to evaluate the presence of reflux in these patients is variable between studies and it seems that this incidence could decrease one year after the procedure.

In recent years, there has been a growing expansion of the application of robot-assisted technology. Robotic Heller myotomy (RHM) has been proposed as an alternative minimally invasive approach to traditional laparoscopy. However, there are doubts regarding the increased cost, longer surgical times, and loss of tactile feedback associated with the robotic approach. A recent systematic review proposes it as an alternative with comparable results to conventional laparoscopy in terms of clinical results and associated morbidity and mortality. Furthermore, it seems that the robotic approach offers a decrease in the rate of mucosal perforation during the procedure that could be related to the greater precision that this technique offers in the dissection of the muscular layer, which ranges between 0-1% and is comparable to that offered by the POEM but lower than the LHM.

Therefore, POEM and RHM could have comparable results in short term, but there is no clear certainty about the results in medium-long term. Likewise, there is a lack of studies that confirm postoperative reflux results in both procedures.

The purpose of the study is evaluate the clinical and quality of life results of RHM and compare them with the results of POEM in the treatment of achalasia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic achalasia with an Eckardt score of > 3 and pre-op barium swallow, manometry and esophagogastroduodenoscopy consistent with the diagnosis
2. Persons of age > 18 years with medical indication for surgical myotomy or EBD
3. Signed written Informed Consent

Exclusion Criteria:

1. Patients with previous surgery of the stomach or esophagus
2. Patients with known coagulopathy
3. Previous myotomy
4. Patients with liver cirrhosis and/or esophageal varices
5. Malignant esophageal lesion
6. Hiatal hernia
7. Extensive dilatation of the esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Eckhard symptom scores | 6 months and 2 years after treatment
  Achalasia symptom questionnaire to evaluate individual therapy success, range from 0 (no Achalasia symptoms) to 12 (full symptom range), treatment success is defined as an Eckardt Score ≤ 3

SECONDARY OUTCOMES:
GERD-Q score | 6 months and 2 years after treatment
  Gastroesophageal reflux questionaire to evaluate individual presence of postreatment reflux, range from 0 (no reflux symptoms) to 18 (full symptom range)

CONTACTS AND LOCATIONS:
Locations (1):
- Elisenda Garsot Savall, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khashab MA, Vela MF, Thosani N, Agrawal D, Buxbaum JL, Abbas Fehmi SM, Fishman DS, Gurudu SR, Jamil LH, Jue TL, Kannadath BS, Law JK, Lee JK, Naveed M, Qumseya BJ, Sawhney MS, Yang J, Wani S. ASGE guideline on the management of achalasia. Gastrointest Endosc. 2020 Feb;91(2):213-227.e6. doi: 10.1016/j.gie.2019.04.231. Epub 2019 Dec 13. PMID 31839408
- [Background] Pandolfino JE, Kwiatek MA, Nealis T, Bulsiewicz W, Post J, Kahrilas PJ. Achalasia: a new clinically relevant classification by high-resolution manometry. Gastroenterology. 2008 Nov;135(5):1526-33. doi: 10.1053/j.gastro.2008.07.022. Epub 2008 Jul 22. PMID 18722376
- [Background] Aiolfi A, Bona D, Riva CG, Micheletto G, Rausa E, Campanelli G, Olmo G, Bonitta G, Bonavina L. Systematic Review and Bayesian Network Meta-Analysis Comparing Laparoscopic Heller Myotomy, Pneumatic Dilatation, and Peroral Endoscopic Myotomy for Esophageal Achalasia. J Laparoendosc Adv Surg Tech A. 2020 Feb;30(2):147-155. doi: 10.1089/lap.2019.0432. Epub 2019 Jul 31. PMID 31364910
- [Background] Zhang H, Zeng X, Huang S, Shi L, Xia H, Jiang J, Ren W, Peng Y, Lu M, Tang X. Mid-Term and Long-Term Outcomes of Peroral Endoscopic Myotomy for the Treatment of Achalasia: A Systematic Review and Meta-Analysis. Dig Dis Sci. 2023 Apr;68(4):1386-1396. doi: 10.1007/s10620-022-07720-4. Epub 2022 Oct 19. PMID 36260203
- [Background] Rohof WO, Salvador R, Annese V, Bruley des Varannes S, Chaussade S, Costantini M, Elizalde JI, Gaudric M, Smout AJ, Tack J, Busch OR, Zaninotto G, Boeckxstaens GE. Outcomes of treatment for achalasia depend on manometric subtype. Gastroenterology. 2013 Apr;144(4):718-25; quiz e13-4. doi: 10.1053/j.gastro.2012.12.027. Epub 2012 Dec 28. PMID 23277105
- [Background] Pratap N, Kalapala R, Darisetty S, Joshi N, Ramchandani M, Banerjee R, Lakhtakia S, Gupta R, Tandan M, Rao GV, Reddy DN. Achalasia cardia subtyping by high-resolution manometry predicts the therapeutic outcome of pneumatic balloon dilatation. J Neurogastroenterol Motil. 2011 Jan;17(1):48-53. doi: 10.5056/jnm.2011.17.1.48. Epub 2011 Jan 26. PMID 21369491
- [Background] Salvador R, Costantini M, Zaninotto G, Morbin T, Rizzetto C, Zanatta L, Ceolin M, Finotti E, Nicoletti L, Da Dalt G, Cavallin F, Ancona E. The preoperative manometric pattern predicts the outcome of surgical treatment for esophageal achalasia. J Gastrointest Surg. 2010 Nov;14(11):1635-45. doi: 10.1007/s11605-010-1318-4. Epub 2010 Sep 10. PMID 20830530
- [Background] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJPM, Pandolfino JE; International Working Group for Disorders of Gastrointestinal Motility and Function. Expert consensus document: Advances in the management of oesophageal motility disorders in the era of high-resolution manometry: a focus on achalasia syndromes. Nat Rev Gastroenterol Hepatol. 2017 Nov;14(11):677-688. doi: 10.1038/nrgastro.2017.132. Epub 2017 Sep 27. PMID 28951579
- [Background] Patel K, Abbassi-Ghadi N, Markar S, Kumar S, Jethwa P, Zaninotto G. Peroral endoscopic myotomy for the treatment of esophageal achalasia: systematic review and pooled analysis. Dis Esophagus. 2016 Oct;29(7):807-819. doi: 10.1111/dote.12387. Epub 2015 Jul 14. PMID 26175119
- [Background] Akintoye E, Kumar N, Obaitan I, Alayo QA, Thompson CC. Peroral endoscopic myotomy: a meta-analysis. Endoscopy. 2016 Dec;48(12):1059-1068. doi: 10.1055/s-0042-114426. Epub 2016 Sep 12. PMID 27617421
- [Background] Werner YB, Hakanson B, Martinek J, Repici A, von Rahden BHA, Bredenoord AJ, Bisschops R, Messmann H, Vollberg MC, Noder T, Kersten JF, Mann O, Izbicki J, Pazdro A, Fumagalli U, Rosati R, Germer CT, Schijven MP, Emmermann A, von Renteln D, Fockens P, Boeckxstaens G, Rosch T. Endoscopic or Surgical Myotomy in Patients with Idiopathic Achalasia. N Engl J Med. 2019 Dec 5;381(23):2219-2229. doi: 10.1056/NEJMoa1905380. PMID 31800987
- [Background] Ponds FA, Fockens P, Lei A, Neuhaus H, Beyna T, Kandler J, Frieling T, Chiu PWY, Wu JCY, Wong VWY, Costamagna G, Familiari P, Kahrilas PJ, Pandolfino JE, Smout AJPM, Bredenoord AJ. Effect of Peroral Endoscopic Myotomy vs Pneumatic Dilation on Symptom Severity and Treatment Outcomes Among Treatment-Naive Patients With Achalasia: A Randomized Clinical Trial. JAMA. 2019 Jul 9;322(2):134-144. doi: 10.1001/jama.2019.8859. PMID 31287522
- [Background] Facciorusso A, Singh S, Abbas Fehmi SM, Annese V, Lipham J, Yadlapati R. Comparative efficacy of first-line therapeutic interventions for achalasia: a systematic review and network meta-analysis. Surg Endosc. 2021 Aug;35(8):4305-4314. doi: 10.1007/s00464-020-07920-x. Epub 2020 Aug 27. PMID 32856150
- [Background] Ciomperlik H, Dhanani NH, Mohr C, Hannon C, Olavarria OA, Holihan JL, Liang MK. Systematic Review of Treatment of Patients with Achalasia: Heller Myotomy, Pneumatic Dilation, and Peroral Endoscopic Myotomy. J Am Coll Surg. 2023 Mar 1;236(3):523-532. doi: 10.1097/XCS.0000000000000484. Epub 2022 Nov 16. PMID 36382896
- [Background] Schlottmann F, Luckett DJ, Fine J, Shaheen NJ, Patti MG. Laparoscopic Heller Myotomy Versus Peroral Endoscopic Myotomy (POEM) for Achalasia: A Systematic Review and Meta-analysis. Ann Surg. 2018 Mar;267(3):451-460. doi: 10.1097/SLA.0000000000002311. PMID 28549006
- [Background] Repici A, Fuccio L, Maselli R, Mazza F, Correale L, Mandolesi D, Bellisario C, Sethi A, Khashab MA, Rosch T, Hassan C. GERD after per-oral endoscopic myotomy as compared with Heller's myotomy with fundoplication: a systematic review with meta-analysis. Gastrointest Endosc. 2018 Apr;87(4):934-943.e18. doi: 10.1016/j.gie.2017.10.022. Epub 2017 Nov 2. PMID 29102729
- [Background] Evensen H, Kristensen V, Larssen L, Sandstad O, Hauge T, Medhus AW. Outcome of peroral endoscopic myotomy (POEM) in treatment-naive patients. A systematic review. Scand J Gastroenterol. 2019 Jan;54(1):1-7. doi: 10.1080/00365521.2018.1549271. Epub 2019 Jan 16. PMID 30650313
- [Background] Khan MA, Kumbhari V, Ngamruengphong S, Ismail A, Chen YI, Chavez YH, Bukhari M, Nollan R, Ismail MK, Onimaru M, Balassone V, Sharata A, Swanstrom L, Inoue H, Repici A, Khashab MA. Is POEM the Answer for Management of Spastic Esophageal Disorders? A Systematic Review and Meta-Analysis. Dig Dis Sci. 2017 Jan;62(1):35-44. doi: 10.1007/s10620-016-4373-1. Epub 2016 Nov 17. PMID 27858325
- [Background] Xie J, Vatsan MS, Gangemi A. Laparoscopic versus robotic-assisted Heller myotomy for the treatment of achalasia: A systematic review with meta-analysis. Int J Med Robot. 2021 Aug;17(4):e2253. doi: 10.1002/rcs.2253. Epub 2021 Apr 12. PMID 33844413
- [Background] Ali AB, Khan NA, Nguyen DT, Chihara R, Chan EY, Graviss EA, Dunkin BJ, Kim MP. Robotic and per-oral endoscopic myotomy have fewer technical complications compared to laparoscopic Heller myotomy. Surg Endosc. 2020 Jul;34(7):3191-3196. doi: 10.1007/s00464-019-07093-2. Epub 2019 Sep 3. PMID 31482358